CLINICAL TRIAL: NCT01407250
Title: Reliability of Outpatient Electrocardiogram Recordings in Patients Refered for a Cardiology Consultation
Brief Title: PhysioGlove Versus Clinic Electrocardiogram Comparison
Acronym: CommwellPG
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Daniel David MD, Commwellmedica Ltd. Israel
Other Study IDs: Commwell PG 101
Record Dates: First submitted 2011-07-24; First posted 2011-08-02 (Estimated); Last update posted 2011-08-02 (Estimated); Status verified 2011-07

CONDITIONS: Patients With Normal ECG; Patients With Pathological ECG

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Comparison of the quality of the outpatient clinic electrocardiogram performed on patients sent to a cardiology consultation with a standard cable and the PhysioGlove-ES electrocardiograms performed in the cardiology clinic.

DETAILED DESCRIPTION:
The correct performance of a 12 lead electrocardiogram depends on the correct placement of the electrocardiogram electrodes in internationally agreed upon anatomic locations on the patient's limbs and chest. This process requires specific training and diligence on the part of the electrocardiogram performer. The literature points towards a progressive quality degradation of the electrocardiogram performance probably due to the delegation of it's performance to lesser trained individuals. This study is attempting to ascertain the quality of the electrocardiogram recordings performed in non-specialized out patient clinics.

For this purpose we will compare outpatient electrocardiograms of patients referred to a cardiological consultation with electrocardiogram's acquired using a conventional electrocardiogram cable as well as the PhysioGlove-ES by the well training cardiology clinic personnel.

ELIGIBILITY:
Inclusion Criteria: all consenting male and female patients age 18-95 -

Exclusion Criteria:

1. All patients using shirt-sizes under small mand over extra-large
2. all patients with severe chest malformations or open wounds or contagious skin infections involving the chest and/or arms -

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult male and female patients
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2011-08; Primary Completion 2011-11 (Estimated); Study Completion 2012-03 (Estimated)

PRIMARY OUTCOMES:
Comparison of the technical and diagnostic quality of outpatient clinic electrocardiogram with the on-site (cardiology consultation clinic) performed electrocardiograms | Each patient will be tested once while visiting the cardiology consultation clinic. No further patient follow-up is planed. Data collection and evaluation is estimated at 6-9 months from study initiation
  The cardiology clinic electrocardiogram will be compared to the out-patient electrocardiogram brought by the patient to the cardiology consultant

CONTACTS AND LOCATIONS:
Locations (1):
- Clalit- Cardiology consult clinic, Netanya, Israel